CLINICAL TRIAL: NCT04585217
Title: A Comparison of the Effect of Suture Material on Blepharoplasty Incision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Michael Yoon, Associate Professor, Oculoplastics, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020P000543
Record Dates: First submitted 2020-10-05; First posted 2020-10-14 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Dermatochalasis; Ptosis, Eyelid
Keywords: Blepharoplasty; Dermatochalasis; Wound healing; Suture; Scar
MeSH Terms: conditions — Cutis Laxa; Blepharoptosis; Cicatrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plain gut suture on right eyelid (Active Comparator): Plain gut suture closure of blepharoplasty incision
  Interventions: Procedure: Randomized laterality of suture materials for closure (6-0 polypropylene monofilament suture vs fast absorbing gut suture on right eyelid)
- Polypropylene suture on right eyelid (Active Comparator): Polypropylene suture closure of blepharoplasty incision
  Interventions: Procedure: Randomized laterality of suture materials for closure (6-0 polypropylene monofilament suture vs fast absorbing gut suture on right eyelid)

INTERVENTIONS:
Procedure: Randomized laterality of suture materials for closure (6-0 polypropylene monofilament suture vs fast absorbing gut suture on right eyelid) — Plain gut suture (6-0 fast absorbing plain gut [Sharpoint "Express gut" TM]) and polypropylene suture (6-0 polypropylene [Ethicon Prolene TM]) will be used to close blepharoplasty incisions. Each patient will have one eyelid using plain gut suture and the other eyelid with polypropylene suture. Each subject will be randomized as to laterality.

SUMMARY:
The objective is to compare the effect of suture material on blepharoplasty incision. Outcomes of blepharoplasty scar and/or cosmesis will be compared between plain gut and polypropylene suture. Additionally, the study will assess whether certain Fitzpatrick skin types are associated with increased rates of poor outcomes after blepharoplasty.

DETAILED DESCRIPTION:
Upper eyelid blepharoplasty is commonly performed surgical procedure. The procedure involves excising excess eyelid skin (sometimes with associated orbicularis oculi muscle and orbital fat). It generally has low risk with high success rate. Although blepharoplasty is usually performed for functional reasons, it can also be performed for purely cosmetic indications. Regardless the indication, patients still expect optimal cosmetic results. Various marking and surgical techniques have been described to maximize functional and aesthetic outcomes. However, there are lacking studies on the optimal suture material for upper blepharoplasty. A comprehensive review of the literature reveals three studies which discuss blepharoplasty outcomes related to suture material. The outcomes of all these studies were heavily influenced by subjective interpretation.

Skin incisions can be closed with adhesives, sutures, staples, or allowed to secondarily granulate. There are many published reports on suture reaction and post-operative results on the face, body, and extremities. However, the eyelid skin is unique - it is the thinnest in the body. Post-operative edema, erythema, cyst and scar formation can have an effect on the cosmetic outcome.

Sutures are the most common method used for closure in this setting. Types of sutures used in clinical practice include absorbable gut and polyglactin and non-absorbable polypropylene, nylon, and polyester. Sutures are most commonly placed as either a continuous running or subcuticular passes with and without reinforcing interrupted sutures. Anecdotally, suture-related complications have been observed in specific racial skin types as well as with various suture materials. Results of this study could lead to a more patient specific blepharoplasty with better and more predictable outcomes therefore improving patient care.

Patients in the outpatient oculoplastics clinic will be evaluated for dermatochalasis and approved for upper blepharoplasty. Enrollment and consent into the study will be performed by the study coordinator. The purpose of the study, risks, benefits, and alternatives will be explained to the patient.

If the patient is interested, he or she will be asked to sign a consent form for both the blepharoplasty procedure and the study. On the day of the procedure, the patient's eyelids and sutures will be randomized. The procedure on each eyelid will performed by the same surgeon.

Patients will have the standard post-operative appointments at 1 week and 3 months. A survey will be given to patients to assess their blepharoplasty scar at each appointment. Deidentified photographs will also be taken of the patients and blindly assessed by the study investigators using an observer scar assessment scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-89 years old
* Patients who qualify for functional blepharoplasty

Exclusion Criteria:

* Patients <18 or >89 years old
* Previous eyelid surgery
* History of connective tissue disease
* Children
* Mental handicap
* Pregnant women
* Incarcerated persons

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Patient Observer Scar Assessment Scale | 3 months
  This validated scale has the patient and observer grade their scar on different components. The observer rates on vascularity, pigmentation, thickness, relief, pliability, surface area, and overall opinion. This is done on a 1 - 10 scale with 1 being completely normal skin and 10 being the worst scar imaginable. The patient rates the scar based on pain, itching, color, stiffness, thickness, irregularity, and overall opinion. This is graded on a 1 - 10 scale with 1 being No (absolutely not) and 10 being Yes (absolutely yes).
  The outcome is a difference of > or = 3-points.

SECONDARY OUTCOMES:
Adverse outcomes per Fitzpatrick skin type | 3 months
  Number and type of adverse outcomes stratified by Fitzpatrick skin type

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Yoon, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

REFERENCES:
- [Background] Jaggi R, Hart R, Taylor SM. Absorbable suture compared with nonabsorbable suture in upper eyelid blepharoplasty closure. Arch Facial Plast Surg. 2009 Sep-Oct;11(5):349-52. doi: 10.1001/archfacial.2009.53. No abstract available. PMID 19797100
- [Background] Scaccia FJ, Hoffman JA, Stepnick DW. Upper eyelid blepharoplasty. A technical comparative analysis. Arch Otolaryngol Head Neck Surg. 1994 Aug;120(8):827-30. doi: 10.1001/archotol.1994.01880320029007. PMID 8049043